CLINICAL TRIAL: NCT04625348
Title: A Multicentre Clinical Test of the Ultracore Repose® Mattress (Frontier Therapeutics Ltd) to Prevent Pressure Ulcers Cat. II-IV in Belgian Nursing Homes
Brief Title: A Multicentre Clinical Test of the Ultracore Repose® Mattress to Prevent Pressure Ulcers Cat. II-IV in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BC-06758
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer; Static air mattress; prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- residents (Experimental): daily care of 40 residents will be provided on the Ultracore Repose® mattress
  Interventions: Device: Ultracore Repose® mattress; Other: experiences and perceptions of healthcare workers

INTERVENTIONS:
Device: Ultracore Repose® mattress — residents will be placed on the Ultracore Repose® mattress for the daily care during 14 days
Other: experiences and perceptions of healthcare workers — Three focus groups will be set- up at the end of the study to provide insights into how caregivers think about the product and to provide a deeper understanding of the difference between the use of the Ultracore Repose® mattress (versus the Repose overlay mattress® and an alternating air mattress)

SUMMARY:
A mixed method desgin study will be conducted to study pressure ulcer incidence Cat. II-IV (including deep- tissue injury,unstageable), not associated with the use of medical devices, on the Ultracore Repose® mattress (Frontier therapeutics Ltd) and to study differences in caretakers' experiences and perceptions when using the Ultracore Repose® mattress versus the Repose overlay mattress®

DETAILED DESCRIPTION:
Quantitative part:

Before the start of the study, nurses on the participating wards will be educated by the researcher about skin observation, pressure ulcer classification, risk assessment, risk assessment, and use of the Ultracore Repose® mattress (Frontier therapeutics Ltd).

Skin assessment and risk assessment are performed on a daily basis by the staff nurses. Reliability testing will be done by the researcher on a weekly basis and without pre-announcement. Reliability checks and compliance with the protocol will be completed by the researcher as well as the collection of additional data.

Qualitative part

Three focus groups will be set- up at the end of the study to provide insights into how caregivers think about the product and to provide a deeper understanding of the difference between the use of the Ultracore Repose® mattress (versus the Repose overlay mattress® and an alternating air mattress).The researcher will encourage group interactions to capture the data and to provide a more comprehensive understanding of experiences and perceptions of using the Ultracore Repose® mattress (versus the Repose overlay mattress® and an alternating air mattress). Non-verbal communication will also be captured in each focus group.

ELIGIBILITY:
Inclusion Criteria:

* High risk of pressure ulcers (Braden score < 12) and/or pressure ulcer category 1
* Bedbound (> 8 hours in bed) or chair bound (> 8 hours in chair)
* Aged > 65 years

Exclusion Criteria:

* Pressure ulcer Category II-IV, deep tissue injury (DTI) or unstageable pressure ulcer
* Expected length of stay < 2 weeks
* End of life care
* Medical contraindication for use of static air support devices

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Incidence rate of pressure ulcers Cat. II-IV | 14 days
  Incidence rate of pressure ulcers Cat. II-IV (including deep- tissue injury, unstageable), not associated with the use of medical devices

SECONDARY OUTCOMES:
caretakers' experiences and perceptions | 7 days
  Insight in caretakers' experiences and perceptions (outcome of the focus group interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Principal Investigator — University Ghent
Locations (5):
- Belgium (5):
  - Bocasa, Heusden-Zolder, Limburg
  - Residentie Kartuizerhof - Vulpia, Lierde, Oost-Vlaanderen
  - Woonzorgcentrum Heilig Hart, Oudenaarde, Oost-Vlaanderen
  - Woonzorgcentrum Egmont, Zottegem, Oost-Vlaanderen
  - Huize Zonnelied, Ieper, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon request
Supporting Information: SAP, CSR
Time Frame: on request